CLINICAL TRIAL: NCT01607580
Title: Risk Stratification-directed Low-dose Glucocorticoid Prophylaxis for Acute GVHD After Unmanipulated Haploidentical Blood and Marrow Transplantation--a Randomized, Controlled, Clinical Trial
Brief Title: Efficacy Study of Low-dose Glucocorticoid Prophylaxis for Acute Graft-versus-host Disease(GVHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, director of Peking University People's Hospital，Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUPH IRB [2012] (26)
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-dose glucocorticoid (Experimental): drug
  Interventions: Drug: low-dose glucocorticoid Methylprednisolone
- no intervention after transplant (Other)
  Interventions: Drug: low-dose glucocorticoid Methylprednisolone

INTERVENTIONS:
Drug: low-dose glucocorticoid Methylprednisolone — patients receive low-dose glucocorticoid from day 5 post transplant
  Other Names: Methylprednisolone

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is one of the best, and sometimes the only, option for the treatment of leukemia. However, GVHD rate was still high after haploidentical HSCT.

It was found in our previous study that CD4/CD8>=1.16、CD56bright NK>1.9×106/kg in the graft was associated with higher risk of developing acute Graft-versus-host Disease (GVHD).

The study hypothesis:

Risk stratification-directed low-dose glucocorticoid prophylaxis for acute GVHD after unmanipulated haploidentical blood and marrow transplantation can reduce the incidence of acute GVHD

DETAILED DESCRIPTION:
patients undergone haploidentical HSCT following day 5 post transplant were randomized to treated group(low-dose glucocorticoid) and controlled group(no intervention).

ELIGIBILITY:
Inclusion Criteria:

* no severe diarrhea no serious infection

Exclusion Criteria:

* serious diarrhea active,uncontrolled infection

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
incidence of acute graft-versus-host disease | paticipants will be followed for the duration of hospital stay,an expected average of 100 days
  number of participants with acute graft-versus-host disease at 100 days

SECONDARY OUTCOMES:
incidence of infection | participants will be followed for the duration of hospital stay,an expected average of 100 days
  number of participants with infection (including bacterium,EB virus, cytomegalovirus and fungus ) at 100 days

OTHER OUTCOMES:
engrafment | participants will be followed for the duration of hospital stay,an expected average of 100 days
  numbers of participants with the engrafment of neutrophilic granulocyte and platelets at 100 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital，Institute of Hematology, Beijing
  - Peking University People's Hospital, Beijing

REFERENCES:
- [Derived] Chang YJ, Xu LP, Wang Y, Zhang XH, Chen H, Chen YH, Wang FR, Han W, Sun YQ, Yan CH, Tang FF, Mo XD, Liu KY, Huang XJ. Effects of Low-Dose Glucocorticoid Prophylaxis on Chronic Graft-versus-Host Disease and Graft-versus-Host Disease-Free, Relapse-Free Survival after Haploidentical Transplantation: Long-Term Follow-Up of a Controlled, Randomized Open-Label Trial. Biol Blood Marrow Transplant. 2019 Mar;25(3):529-537. doi: 10.1016/j.bbmt.2018.11.020. Epub 2018 Nov 24. PMID 30481596
- See also: hospital website — http://www.phbjmu.edu.cn